CLINICAL TRIAL: NCT01449799
Title: A Randomised, Double-blind, Double-dummy, Single Dose, Four Way Cross-over Study to Compare the Pharmacokinetics and Pharmacodynamics of GSK961081 and Fluticasone Propionate When Administered Alone, Concurrently and as a Combination Blend in Healthy Subjects
Brief Title: An Investigation of the Pharmacokinetics of GSK961081 and Fluticasone Propionate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113423
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): In period 1, subjects will be administered GSK961081/fluticasone propionate blend via Diskus inhaler followed by the administration of GSK961081 and fluticasone propionate concurrently via separate Diskus inhalers in period 2. In period 3 and period 4, the subjects will receive fluticasone propionate and GSK961081 respectively.
  Interventions: Drug: GSK961081 800 microgram dose; Drug: Fluticasone Propionate 500 microgram dose; Drug: GSK961081 800 microgram and Fluticasone Propionate 500 microgram separately; Drug: GSK961081 800 microgram Fluticasone Propionate 500 microgram in a blend
- Sequence 2 (Experimental): In period 1, subjects will be administered GSK961081 and fluticasone propionate concurrently via separate Diskus inhalers followed by administration of GSK961081 in period 2. In period 3 and period 4, the subjects will receive GSK961081/fluticasone propionate blend via Diskus inhaler followed by the administration of fluticasone propionate respectively.
  Interventions: Drug: GSK961081 800 microgram dose; Drug: Fluticasone Propionate 500 microgram dose; Drug: GSK961081 800 microgram and Fluticasone Propionate 500 microgram separately; Drug: GSK961081 800 microgram Fluticasone Propionate 500 microgram in a blend
- Sequence 3 (Experimental): In period 1, subjects will be administered GSK961081 followed by administration of fluticasone propionate in period 2. In period 3, subjects will be administered GSK961081 and fluticasone propionate concurrently via separate Diskus inhalers followed by GSK961081/fluticasone propionate blend via Diskus inhaler in period 4.
  Interventions: Drug: GSK961081 800 microgram dose; Drug: Fluticasone Propionate 500 microgram dose; Drug: GSK961081 800 microgram and Fluticasone Propionate 500 microgram separately; Drug: GSK961081 800 microgram Fluticasone Propionate 500 microgram in a blend
- Sequence 4 (Experimental): In period 1, subjects will be administered fluticasone propionate followed by the administration of GSK961081/fluticasone propionate blend via Diskus inhaler in period 2. The subjects will receive GSK961081 in period 3 and concurrent administration of GSK961081 and fluticasone propionate in period 4.
  Interventions: Drug: GSK961081 800 microgram dose; Drug: Fluticasone Propionate 500 microgram dose; Drug: GSK961081 800 microgram and Fluticasone Propionate 500 microgram separately; Drug: GSK961081 800 microgram Fluticasone Propionate 500 microgram in a blend

INTERVENTIONS:
Drug: GSK961081 800 microgram dose — To be provided via a combination of 4 inhalers - one 400 micrograms GSK961081 Diskus inhalation, a second 400 microgram GSK961081 Diskus inhalation and one inhalation each from two separate placebo Diskus inhalers
Drug: Fluticasone Propionate 500 microgram dose — To be provided via a combination of 4 inhalers - one 250 microgram fluticasone propionate Diskus inhalation, a second 250 microgram fluticasone proopionate Diskus inhalation, and one inhalation each from two separate placebo Diskus inhalers
Drug: GSK961081 800 microgram and Fluticasone Propionate 500 microgram separately — To be provided via a combination of 4 inhalers - one 400 microgram GSK961081 Diskus inhalation, a second 400 microgram GSK961081 Diskus inhalation, one 250 microgram fluticasone propionate Diskus inhalation, and a second fluticasone propionate 250 microgram Diskus inhalation
Drug: GSK961081 800 microgram Fluticasone Propionate 500 microgram in a blend — To be provided via a combination of 4 inhalers - one inhalation of a Diskus inhaler containing a blend of 400 microgram of GSK961081 and 250 microgram of fluticasone propionate per inhalation, a second inhalation of a Diskus inhaler containing a blend of 400 microgram of GSK961081 and 250 microgram of fluticasone propionate per inhalation, and one inhalation each from two separate placebo inhalers

SUMMARY:
In the current study GSK961081 and fluticasone propionate will be administered in a blended formulation from a single device and compared with GSK961081 and fluticasone propionate administered alone and concurrently. This is a single centre, randomized, double-blind, double dummy, single dose, four way cross-over study investigating the pharmacokinetics and pharmacodynamics of GSK961081 and fluticasone propionate when administered alone, concurrently and as a combination blend in healthy subjects.

DETAILED DESCRIPTION:
This will be the first time that GSK961081 and fluticasone propionate will be administered as a blend in humans. In previous clinical studies conducted in Chronic Obstructive Pulmonary Disease (COPD) patients, GSK961081 has been administered on a background of fluticasone propionate without any observed systemic pharmacodynamic interaction. In this study GSK961081 and fluticasone propionate will be administered in a blended formulation from a single device and compared with GSK961081 and fluticasone propionate administered alone and concurrently. The aim of the study will be to investigate any differences in pharmacodynamics and/or pharmacokinetics for GSK961081 and fluticasone propionate when administered as the blend, concurrently or alone.

Pharmacokinetic, pharmacodynamic and safety information will be gathered to assess the suitability of the GSK9610981/fluticasone propionate blend for further development.Each subject will receive four treatments (GSK961081 alone, fluticasone propionate alone, GSK961081 and fluticasone propionate concurrently, and GSK961081/fluticasone propionate blend) in randomized order, in four treatment periods, each separated by a washout period of at least a week. All treatments will be administered via a DISKUS inhaler.

Pharmacokinetics, pharmacodynamics and safety will be assessed by measurement of plasma GSK961081, plasma fluticasone propionate, serum cortisol, urine cortisol, blood glucose, serum potassium, Forced Expiratory Volume in one second (FEV1), heart rate, 12-lead Electrocardiograms (ECGs), clinical laboratory tests and collection of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
2. Healthy as determined by the Investigator based on a medical evaluation including medical history, physical examination, laboratory tests and lung function testing. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and outcome.
3. A female subject of child bearing potential, is eligible if she agrees to use one of the contraception methods listed in Section 8.1 of the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for 5 half-lives after the end of the study (i.e. until after the follow-up visit is complete).
4. Body Mass Index (BMI) within the range 19.0 - 29.9 kilogram per square meter (kg/m2) (inclusive).
5. Aspartate Transaminase (AST), Alanine Transaminase (ALT), alkaline phosphatase and bilirubin less than 1.5 times the upper limit of normal (<1.5xULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is less than 35%).
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. Forced Expiratory Volume in 1 second (FEV1) greater than or equal to 80% predicted and a FEV1/ Forced Vital Capacity (FVC) ratio greater than or equal to 0.7.
8. Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of less than or equal to 10 pack years.

[number of pack years = (number of cigarettes per day/20) x number of years smoked]

Exclusion Criteria:

1. Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or electrocardiogram (ECG, 12-lead)
2. History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (around 240 millilitres, ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
3. QTc value corrected for Bassett or Fredericia [QTc(B) and QTc(F)] at screening greater than 450 milliseconds on an individual ECG, the 3 screening ECGs are not within 10% of the mean QTC value, a PR interval outside the range 120-210 msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T wave).
4. A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
5. A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
6. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
7. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
8. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
9. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
10. Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 90 day period.
11. Pregnant females as determined by positive serum Human Chorionic Gonadotrophin (hCG test) at screening or prior to dosing.
12. Lactating females.
13. Unwillingness or inability to follow the procedures outlined in the protocol.
14. Subject is mentally or legally incapacitated.
15. A history of respiratory disease (i.e. history of asthmatic symptoms) in the last 10 years.
16. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
17. A positive test for human immunodeficiency virus (HIV) antibody.
18. Urinary Cotinine/ Breath carbon monoxide (CO) levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
19. Night shift workers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07-13 (Actual); Primary Completion 2011-09-21 (Actual); Study Completion 2011-09-21 (Actual)

PRIMARY OUTCOMES:
Plamsa concentrations and derived pharmacokinetic parameters of GSK961081 and fluticasone propionate | From dosing to 24 hours post-dose
  Maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve, and apparent terminal phase half-life (t1/2)] for GSK961081 and fluticasone propionate

SECONDARY OUTCOMES:
Serum Cortisol | From dosing to 24 hours post-dose
  Concentration of the hormone cortisol in serum
Urinary Cortisol | From dosing to 24 hours post-dose
  Concentration of the hormone cortisol in urine
Heart Rate Changes | From dosing to 4 hours post-dose
  The maximum change and weighted mean change in heart rate from baseline (pre-dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Norris V, Ambery C, Riley T. Pharmacokinetics and pharmacodynamics of GSK961081, a novel inhaled muscarinic antagonist beta2 -agonist, and fluticasone propionate administered alone, concurrently and as a combination blend formulation in healthy volunteers. Clin Pharmacol Drug Dev. 2014 Jul;3(4):305-13. doi: 10.1002/cpdd.105. Epub 2014 Feb 20. PMID 27128837
- See also: Results for study 113423 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113423?search=study&search_terms=113423#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113423 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register